CLINICAL TRIAL: NCT01249274
Title: Progesterone for Postpartum Cocaine Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kimberly Yonkers, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1005006793; R21DA029914 (NIH)
Record Dates: First submitted 2010-11-22; First posted 2010-11-29 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Cocaine Abuse; Cocaine Dependence
Keywords: cocaine abuse; cocaine dependence; postpartum period
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matched placebo pills to be taken twice daily
  Interventions: Other: Placebo
- Progesterone (Experimental): 100 mgs progesterone twice daily
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — 100mgs progesterone twice daily
  Other Names: prometrium
  Arms: Progesterone
Other: Placebo — Matched placebo pills to be taken twice daily
  Arms: Placebo

SUMMARY:
The investigators propose a placebo-controlled, randomized clinical trial that would enroll 50 postpartum women with a history of cocaine abuse or dependence to assess whether progesterone (100mgs twice daily) decreases postpartum cocaine use.

DETAILED DESCRIPTION:
Specific Aim 1: To evaluate whether postpartum women with a history of cocaine abuse or dependence use less cocaine if they are randomized to progesterone than placebo.

Hypothesis 1: Compared to women who are randomized to placebo, those assigned to progesterone will use less cocaine as measured by urine toxicology results and self-reported days of use.

Specific aim 2: To obtain information about the safety and tolerability of progesterone treatment in the postpartum period.

Hypothesis 2: Side effects for progesterone will be similar to those of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Gravidas (women who delivered a baby in the past 12 weeks) who are 18 or older are eligible to participate.
* Women must meet diagnostic criteria for abuse or dependence of cocaine in the six-months prior to conception or during pregnancy.
* Women who abuse other illicit substances or alcohol would also be eligible as long as cocaine was their primary drug of abuse. If women are also opiate dependent, they must be undergoing treatment with methadone or buprenorphine. While we propose to target cocaine we will also monitor the ability of women with polysubstance use to maintain abstinence from substances other than cocaine.

Exclusion Criteria:

Women will be ineligible for the trial if they:

1. have a history of major medical illnesses including liver diseases, suspected or known malignancy, thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders, heart disease, diabetes, history of stroke or other medical conditions that the physician investigator deems as contraindicated for participation in the study;
2. have a known allergy to progesterone or peanuts (vehicle for micronized progesterone);
3. speak a language other than English;
4. are planning on moving out of the area in the first six months after delivery;
5. are unable to understand the study or are unable to provide informed consent;
6. are currently undergoing treatment with another pharmacological agent for substance abuse treatment (with the exception of methadone or buprenorphine as above);
7. have pending incarceration;
8. are currently incarcerated;
9. are using another progestin;
10. are unwilling to accept randomization;
11. are unwilling to use a barrier method of birth control for the duration of the study to ensure that they will not become pregnant.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Yonkers, MD, Principal Investigator — Yale University; Mehmet Sofuoglu, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Data request should be made to the PI

REFERENCES:
- See also: Research site webpage — http://researchforher.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On-site clinic screening assessments were performed in three obstetrics clinic associated with the Yale New Haven Hospital System in New Haven, CT, USA. Study referrals were accepted from the New Haven area. Both post-partum and pregnant women were screened. Screenings began in October of 2010 and finished in February of 2013.
Pre-assignment Details: 75 women were scheduled for intake, but 24 did not complete intake interview and 1 was ineligible for randomisation because of a medical issue. The first 50 eligible women were randomly assigned.
Period: Overall Study
Arm/Group | Placebo | Progesterone
Started | 25 (all 25 were included in intention-to-treat and safety analyses) | 25 (all 25 were included in intention-to-treat and safety analyses)
Completed Treatment | 21 | 19
Completed Treatment & Post Trial Visit | 20 | 17
Completed Post Trial Visit But Not tx | 1 | 2
Completed | 21 | 19
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 3 | 4
Not completed — Received inpatient substance treatment | 1 | 2

BASELINE CHARACTERISTICS:
Population: All 25 in each study group were included in intention-to-treat and safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Progesterone | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (6.3) | 30.5 (4.5) | 31.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 16 | 28
  Black | 12 | 4 | 16
  Hispanic or other | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Education [Number; unit: participants]
  Less than high shool | 9 | 4 | 13
  High school | 8 | 9 | 17
  Post-high school | 8 | 12 | 20
Marital status [Number; unit: participants]
  Married or cohabitating | 5 | 7 | 12
  Divorced | 3 | 1 | 4
  Separated | 2 | 2 | 4
  Dating | 6 | 1 | 7
  Single | 9 | 14 | 23
Employment status [Number; unit: participants]
  In paid employment | 7 | 3 | 10
  Not in paid employment | 17 | 20 | 37
  Unknown | 1 | 2 | 3
Weeks post partum [Mean (Standard Deviation); unit: weeks] | 3.4 (5.1) | 3.6 (4.6) | 3.5 (2.3)
Lifetime cocaine use (years) [Mean (Standard Deviation); unit: years] | 8.5 (7.2) | 6.2 (4.2) | 7.4 (2.8)
Age at first cocaine use (years) [Mean (Standard Deviation); unit: years] | 20.6 (6.3) | 19.2 (4.0) | 19.9 (2.2)
Parity [Mean (Standard Deviation); unit: births] | 2.6 (1.6) | 2.1 (1.4) | 2.4 (0.2)
EPDS score at intake [Mean (Standard Deviation); unit: units on a scale] — The Edinburgh Postnatal Depression scale measures depression and has 10 items with range of 0-30. Higher scores indicate more severe depression.
  units on a scale | 11.2 (6.7) | 11.2 (7.2) | 11.2 (3.9)
Baseline cocaine use (days per week) [Mean (Standard Deviation); unit: days] — Baseline cocaine use (days of use per week, averaged across 4 weeks prior to baseline, maximum value=7 days)
  days | 0.41 (.91) | 1.15 (3.84) | 1.1 (1.0)
Not using cocaine at intake [Number; unit: participants]
  Not using cocaine at intake | 22 | 19 | 41
  Using cocaine at intake | 3 | 6 | 9
Methadone maintained [Number; unit: participants]
  Using methadone | 8 | 14 | 22
  not using methadone | 17 | 11 | 28
Any lifetime major depressive episode [Number; unit: participants]
  History of MDD | 4 | 3 | 7
  No history of MDD | 21 | 22 | 43
Social phobia [Number; unit: participants]
  History of social phobia | 5 | 1 | 6
  No history of social phobia | 20 | 24 | 44
Obsessive compulsive disorder [Number; unit: participants]
  yes | 4 | 0 | 4
  no | 21 | 25 | 46
Generalized anxiety disorder [Number; unit: participants]
  yes | 6 | 8 | 14
  no | 19 | 17 | 36
Post-traumatic stress disorder [Number; unit: participants]
  yes | 5 | 6 | 11
  no | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Days Per Week of Cocaine Use
Description: Primary aim: to evaluate whether postpartum women with a history of cocaine abuse or dependence use less cocaine if they are randomized to progesterone than placebo. Measured by self-reported days of cocaine use per week via substance use calendar.
Time Frame: Weekly measurements, Baseline to 12 weeks
Population: intent-to-treat
Measure: Mean (Standard Deviation); unit: number of days per week of cocaine use
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
number of days per week of cocaine use
  Baseline | 0.41 (0.91) | 1.15 (3.84)
  Week 1 | 0.43 (0.88) | 1.01 (3.15)
  Week 2 | 0.45 (0.89) | 0.89 (2.51)
  Week 3 | 0.47 (0.91) | 0.78 (2.16)
  Week 4 | 0.49 (0.94) | 0.68 (1.87)
  Week 5 | 0.52 (1.02) | 0.60 (1.62)
  Week 6 | 0.52 (1.13) | 0.53 (1.41)
  Week 7 | 0.56 (1.30) | 0.46 (1.18)
  Week 8 | 0.59 (1.37) | 0.41 (1.04)
  Week 9 | 0.62 (1.55) | 0.36 (0.92)
  Week 10 | 0.64 (1.68) | 0.31 (0.89)
  Week 11 | 0.67 (1.91) | 0.28 (0.76)
  Week 12 | 0.70 (2.11) | 0.24 (0.68)
Statistical Analysis 1: Comparison: Placebo vs Progesterone; Test type: Superiority or Other; p = 0.010, Generalized Estimating Equation; Negative binomial distribution, log link, and first-order autoregressive covariance structure; Risk Ratio (RR) = 1.19, 95% CI 2-sided [1.04 to 1.36] — Estimated value is the risk ratio estimate for the treatment x time interaction term. Time was treated as a continuous variable and progesterone was the reference group for the treatment variable

2. Primary Outcome: Number of Days of Cocaine Use Between 12 Week Visits & the 3 Month Follow up
Description: Primary aim: to evaluate whether postpartum women with a history of cocaine abuse or dependence use less cocaine if they are randomized to progesterone than placebo. Measured by self-reported days of cocaine use per week during the trial period and during 3 month follow up using the substance use calendar
Time Frame: baseline, end of trial (week 12), 3-month post-trial follow-up
Population: intent-to-treat
Measure: Mean (95% Confidence Interval); unit: days of cocaine use between visits
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
days of cocaine use between visits
  Baseline | 0.5200 [0.1419 to 1.9062] | 1.6800 [0.5983 to 4.7171]
  End of Trial (Week 12) | 0.2860 [0.1237 to 0.6609] | 0.05550 [0.009978 to 0.3087]
  3-Month Post-Trial Follow-Up | 12.8472 [5.3751 to 30.7066] | 1.3659 [0.2618 to 7.1263]
Statistical Analysis 1: Comparison: Placebo vs Progesterone; We calculated that a sample size of 50 women would have 80% power to detect a significant (p<0.05) difference between groups if the effect size for the primary outcome was large; Test type: Superiority or Other; p = 0.003, Generalized Estimating Equation; Negative binomial distribution, log link, and first-order autoregressive covariance structure; Risk Ratio (RR) = 30.39, 95% CI 2-sided [3.18 to 290.04] — Estimated value is RR for treatment*time interaction for placebo at 3-mo post-trial follow-up. Time treated as a 3-level categorical variable; week 0 (ref), week 12 & 3-month post-trial follow-up. Treatment variable reference group was progesterone
Statistical Analysis 2: Comparison: Placebo vs Progesterone; Negative binomial distribution, log link, and first-order autoregressive covariance structure; Test type: Superiority or Other; p = 0.038, Generalized Estimating Equation; Risk Ratio (RR) = 16.65, 95% CI 2-sided [1.18 to 235.52] — Estimated value is RR for treatment*time interaction term for placebo at week 12. Time was treated as a 3-level categorical variable; week 0 (ref), week 12 and 3-month post-trial follow-up. Treatment variable reference group was progesterone

3. Primary Outcome: Proportion of Positive Urine Samples Per Week
Description: Primary aim: to evaluate whether postpartum women with a history of cocaine abuse or dependence use less cocaine if they are randomized to progesterone than placebo. Urine tox tests obtained qualitative and quantitative data on cocaine metabolites and other substances.
Time Frame: weekly measurements, baseline to 12 weeks
Population: intent-to-treat
Measure: Mean (95% Confidence Interval); unit: proportion of positive urines per week
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
proportion of positive urines per week
  Baseline | 0.2645 [0.1278 to 0.4688] | 0.1990 [0.0882 to 0.3893]
  Week 1 | 0.2667 [0.1366 to 0.4554] | 0.2006 [0.0928 to 0.3810]
  Week 2 | 0.2689 [0.1448 to 0.4443] | 0.2022 [0.0969 to 0.3745]
  Week 3 | 0.2712 [0.1519 to 0.4360] | 0.2038 [0.1003 to 0.3702]
  Week 4 | 0.2734 [0.1576 to 0.4309] | 0.2054 [0.1029 to 0.3681]
  Week 5 | 0.2757 [0.1613 to 0.4296] | 0.2071 [0.1047 to 0.3685]
  Week 6 | 0.2780 [0.1629 to 0.4323] | 0.2087 [0.1054 to 0.3714]
  Week 7 | 0.2803 [0.1623 to 0.4390] | 0.2104 [0.1051 to 0.3768]
  Week 8 | 0.2826 [0.1597 to 0.4494] | 0.2121 [0.1038 to 0.3847]
  Week 9 | 0.2849 [0.1553 to 0.4633] | 0.2138 [0.1017 to 0.3949]
  Week 10 | 0.2872 [0.1496 to 0.4799] | 0.2154 [0.0989 to 0.4071]
  Week 11 | 0.2895 [0.1429 to 0.4989] | 0.2171 [0.0956 to 0.4213]
  Week 12 | 0.2918 [0.1356 to 0.5198] | 0.2189 [0.0918 to 0.4372]
Statistical Analysis 1: Comparison: Placebo vs Progesterone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.99, Generalized Estimating Equation; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.87 to 1.15] — Estimated value is the risk ratio for the treatment x time interaction term. Time was treated as a continuous variable and progesterone was the reference group for treatment

4. Primary Outcome: Proportion of Positive Urine Samples Per Week
Description: as for outcome 3
Time Frame: baseline, end of trial (week 12) and 3-month post-trial follow-up
Population: intent-to-treat
Measure: Mean (95% Confidence Interval); unit: proportion of positive urines per week
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
proportion of positive urines per week
  Baseline | 0.2400 [0.1120 to 0.4416] | 0.1582 [0.0559 to 0.3733]
  Week 12 | 0.3173 [0.1606 to 0.5303] | 0.1904 [0.0758 to 0.4028]
  3 month post-trial follow-up | 0.3952 [0.2189 to 0.6037] | 0.2246 [0.0852 to 0.4740]
Statistical Analysis 1: Comparison: Placebo vs Progesterone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.75, Generalized Estimating Equation; Risk Ratio (RR) = 1.34, 95% CI 2-sided [0.23 to 7.88] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Progesterone; Test type: Superiority or Other; p = 0.84, Generalized Estimating Equation; Negative binomial distribution, log link, and first-order autoregressive covariance structure; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.24 to 5.84] — Estimated value is RR for treatment*time interaction for placebo at week 12. Time was treated as a 3-level categorical variable; week 0 (ref), week 12 & 3-month post-trial follow-up. Treatment variable reference group was progesterone

5. Secondary Outcome: Overall Comparison of Adverse Events Between Women in Placebo and Progesterone Group
Description: To obtain information about the safety and tolerability of progesterone treatment in the postpartum period, women were queried at every visit about onset of adverse events, their seriousness, and their relatedness to study medication. Such data was monitored in SAETRS.
Time Frame: 12 weeks postpartum
Population: intent-to-treat
Measure: Number; unit: adverse events
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
adverse events | 11 | 15
Statistical Analysis 1: Comparison: Placebo vs Progesterone; Test type: Superiority or Other; p = 0.1030, Fisher Exact

6. Secondary Outcome: Cocaine Craving (Measured Weekly Using CCQ-Brief)
Description: CCQ-Brief is a ten-item questionnaire developed from the 45-item CCQ. Each item is scored on a visual analogue scale ranging from 1-7, and items are averaged to yield a score from 1 to 7. Higher scores indicate stronger cocaine cravings.
Time Frame: baseline to 12 weeks
Population: intent-to-treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 1.5630 [1.2953 to 1.8860] | 1.6752 [1.3609 to 2.0620]
  Week 1 | 1.5456 [1.3073 to 1.8275] | 1.6532 [1.3616 to 2.0073]
  Week 2 | 1.5285 [1.3161 to 1.7751] | 1.6316 [1.3594 to 1.9583]
  Week 3 | 1.5115 [1.3205 to 1.7301] | 1.6102 [1.3536 to 1.9154]
  Week 4 | 1.4947 [1.3189 to 1.6939] | 1.5891 [1.3438 to 1.8791]
  Week 5 | 1.4781 [1.3097 to 1.6681] | 1.5683 [1.3297 to 1.8497]
  Week 6 | 1.4616 [1.2925 to 1.6530] | 1.5478 [1.3111 to 1.8271]
  Week 7 | 1.4454 [1.2678 to 1.6478] | 1.5275 [1.2883 to 1.8111]
  Week 8 | 1.4293 [1.2374 to 1.6510] | 1.5075 [1.2619 to 1.8009]
  Week 9 | 1.4134 [1.2032 to 1.6604] | 1.4877 [1.2325 to 1.7957]
  Week 10 | 1.3977 [1.1668 to 1.6744] | 1.4682 [1.2010 to 1.7949]
  Week 11 | 1.3822 [1.1292 to 1.6919] | 1.4490 [1.1681 to 1.7975]
  Week 12 | 1.3668 [1.0914 to 1.7118] | 1.4300 [1.1342 to 1.8030]
Statistical Analysis 1: Comparison: Placebo vs Progesterone; Test type: Superiority or Other; p = 0.9116, Generalized Estimating Equation; Gamma distribution, logit link, 1st-order autoregressive covariance structure; p-value is for chi-sq (df=1) for type 3 GEE analysis score statistic; Score Statistic For Type 3 GEE Analysis = 0.01 — Estimated value is chi-sq (df=1) for type 3 GEE analysis score statistic for week*treatment interaction term

7. Secondary Outcome: Depression (Measured Weekly Using Edinburgh Postnatal Depression Scale (EPDS))
Description: EPDS scores were measured to detect depression as a possible adverse event and compare scores between the two groups. The scale consists of 10 items. Each item is scored from 0 to 3, and the 10 items are summed to calculate a total score with a possible range of 0 to 30 and higher scores indicating more severe depression.
Time Frame: baseline to 12 weeks
Population: intent-to-treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
units on a scale
  Baseline | 10.84 (1.37) | 11.08 (1.44)
  Week 1 | 8.05 (1.37) | 8.61 (1.41)
  Week 2 | 8.57 (1.19) | 6.65 (1.03)
  Week 3 | 6.91 (1.04) | 6.95 (1.41)
  Week 4 | 9.27 (1.60) | 6.62 (1.08)
  Week 5 | 7.60 (1.54) | 6.62 (1.09)
  Week 6 | 8.05 (1.52) | 7.24 (1.48)
  Week 7 | 9.13 (1.71) | 6.53 (1.41)
  Week 8 | 8.29 (1.64) | 6.16 (1.48)
  Week 9 | 8.24 (1.70) | 6.68 (1.77)
  Week 10 | 8.55 (1.69) | 6.64 (1.33)
  Week 11 | 7.33 (1.43) | 6.85 (1.40)
  Week 12 | 8.38 (1.71) | 6.60 (1.15)
  3-month post trial | 9.09 (1.43) | 7.21 (1.32)

8. Secondary Outcome: Salivary Progesterone Concentrations
Description: A comparison of salivary progesterone concentrations across all samples for all timepoints
Time Frame: week 2, week 6, week 10, week 12
Population: intent-to-treat
Measure: Mean (Standard Error); unit: pg/ml of salivary progesterone
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 25 | 25
pg/ml of salivary progesterone
  Week 2 | 165.94 (135.30) | 797.26 (1004.13)
  Week 6 | 189.38 (237.94) | 1580.95 (1963.51)
  Week 10 | 124.30 (72.31) | 1771.07 (3139.36)
  Week 12 | 235.04 (288.51) | 866.10 (1044.84)

9. Post Hoc Outcome: Relapse to Cocaine Use During Treatment Period
Description: Post-hoc sensitivity test to compare hazard of relapse to cocaine use between two treatment groups among participants (n=41) who did not report using cocaine at intake.
Time Frame: baseline to 12 weeks
Population: intent-to-treat
Measure: Number; unit: participants who relapsed to cocaine use
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 22 | 19
participants who relapsed to cocaine use | 9 | 3
Statistical Analysis 1: Comparison: Placebo vs Progesterone; Test type: Superiority or Other; p = 0.048, Regression, Cox; Cox Proportional Hazard = 4.71, 95% CI 2-sided [1.09 to 20.50] — Ratio presented is for placebo versus progesterone

10. Post Hoc Outcome: Relapse to Cocaine Use During Treatment Period or 3 Months Post Treatment
Description: as for outcome 9
Time Frame: baseline to 3 months post 12-week trial period
Population: intent-to-treat
Measure: Number; unit: participants who relapsed to cocaine use
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 22 | 19
participants who relapsed to cocaine use | 10 | 4
Statistical Analysis 1: Comparison: Placebo vs Progesterone; Test type: Superiority or Other; p = 0.06, Regression, Cox; Cox Proportional Hazard = 3.50, 95% CI 2-sided [0.92 to 13.30] — Ratio presented is for placebo versus progesterone

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the entire study period, from the intake of the participants to their final 3-month follow-up.
Arm/Group | Placebo | Progesterone
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 11/25 | 15/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Progesterone (N=25)
Headache (General disorders) | 3 (3) | 6 (6)
Sedation (General disorders) | 4 (4) | 4 (4)
Dizziness (General disorders) | 0 (0) | 3 (3)
Dry mouth (General disorders) | 3 (3) | 0 (0)
Nausea (General disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Women seen only once per week leading to reliance on self-reports more than urine, results of which differed; post-partum women with cocaine use disorder have other issues affecting likelihood of cocaine use; missed visits may have biased results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No